CLINICAL TRIAL: NCT07198126
Title: Comparison Of Keratometric Readings Pre and Post Pterygium Excision With Conjunctival Autograft Transplantation
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Mughal Eye Trust Hospital (Other)
Responsible Party: Principal Investigator, Ayeza Nadeem Butt, Principal Investigator, Mughal Eye Trust Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MughalETH1
Record Dates: First submitted 2025-09-21; First posted 2025-09-30 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Pterygium; Corneal Astigmatism
Keywords: Pterygium excision; Astigmatism correction; Conjunctival autograft transplantation; Refractive error
MeSH Terms: conditions — Pterygium; Astigmatism; Refractive Errors

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Group Pterygium Excision with Conjunctival Autograft (Experimental): Patients will undergo surgical excision of pterygium followed by conjunctival autograft transplantation. The autograft will be harvested from the superior bulbar conjunctiva and secured at the excision site using sutures.
  Interventions: Procedure: Pterygium Excision with Conjunctival Autograft

INTERVENTIONS:
Procedure: Pterygium Excision with Conjunctival Autograft — Excision of primary Grade II or Grade III pterygium Conjunctival autograft harvested and transplanted at the excision site Graft secured with sutures

SUMMARY:
Pterygium, often called "surfer's eye," is a common eye condition in which a raised, fleshy growth of tissue extends from the white part of the eye onto the clear cornea. This growth can cause redness, irritation, blurred vision, and, in advanced cases, changes in the curvature of the cornea leading to distorted vision (astigmatism). The condition is more frequent in people exposed to sunlight, dust, and dry environments.

The standard treatment for symptomatic pterygium is surgical removal. However, simple removal has a high chance of recurrence. To reduce this risk, surgeons commonly use a technique called conjunctival autograft transplantation, where a small piece of the patient's own conjunctiva is placed over the area after excision. This method not only lowers the recurrence rate but may also improve vision by reducing corneal irregularities.

This study is designed to measure the changes in corneal curvature (keratometric readings) before and after pterygium excision with conjunctival autograft transplantation. By comparing preoperative and postoperative measurements, the study aims to determine how much this surgery improves corneal shape and reduces astigmatism.

The hypothesis is that pterygium excision with conjunctival autograft transplantation will lead to a significant improvement in keratometric readings and reduce irregular astigmatism, thereby improving visual quality.

This research will provide local evidence of the effectiveness of this procedure and help guide treatment strategies for patients suffering from pterygium-related visual problems.

ELIGIBILITY:
Inclusion Criteria:

* Adults of either sex aged >30 to 70 years.
* Phakic eyes.
* Primary pterygium, Grade II or Grade III (as per protocol grading).
* Presence of corneal astigmatism on pre-operative assessment.
* Scheduled for pterygium excision with conjunctival autograft transplantation at the study site.
* Able to provide written informed consent and to attend the 1-month postoperative assessment.

Exclusion Criteria:

* Pseudophakic or aphakic eyes.
* Recurrent pterygium.
* Prior keratoplasty or trabeculectomy in the study eye.
* Keratoconus or other corneal pathologies that can independently induce astigmatism.
* Lenticular astigmatism or significant lens pathology affecting refraction.
* Eyes planned for simple pterygium excision without conjunctival autograft.
* Any ocular condition or systemic illness judged likely to interfere with keratometric or refractive measurements, follow-up, or surgical safety.

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2025-08-30 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Change in Keratometric Readings (K1 and K2) | Baseline (pre-operative) and 1 month post-operative.
  Keratometric readings, including the flat meridian (K1) and steep meridian (K2) of the anterior corneal surface, will be measured using a manual keratometer. The mean change in K-readings (measured in diopters) from baseline (pre-operative) to post-operative assessment will be calculated to evaluate corneal curvature improvement following pterygium excision with conjunctival autograft.

SECONDARY OUTCOMES:
Change in Astigmatism | Baseline (pre-operative) and 1 month post-operative.
  Astigmatism will be measured using an automated refractometer. Both type (regular/irregular, with-the-rule/against-the-rule) and degree of astigmatism (in diopters) will be recorded. The reduction in astigmatism from baseline to post-operative follow-up will be assessed.

CONTACTS AND LOCATIONS:
Locations (1):
- Mughal Eye Hospital Trust, Lahore, Punjab Province, Pakistan